CLINICAL TRIAL: NCT02618044
Title: Long Term Effects of Laparoscopic Roux-en-Y Gastric Bypass on Gastro-esophageal Reflux: Clinical Impact of Weakly Acidic Reflux
Brief Title: Laparoscopic Roux-en-Y Gastric Bypass and Gastro-esophageal Reflux
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Fabrizio Rebecchi, MD, University of Turin, Italy
Other Study IDs: WAROB/97
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Gastroesophageal Reflux; Obesity
Keywords: Gastroesophageal reflux; Obesity; Esophageal manometry; 24 H impedance pH-monitoring; Laparoscopic Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese patients without preoperative GER: Obese patients selected for laparoscopic Roux-en-Y Gastric Bypass without preoperative GER at 24h-impedance pH monitoring (Group G-)
- Obese patients with preoperative GER: Obese patients selected for laparoscopic Roux-en-Y Gastric Bypass with preoperative GER at 24h-impedance pH monitoring (Group G+)

SUMMARY:
Laparoscopic Roux-en-Y Gastric Bypass (LRYGB) is considered the weight loss procedure of choice for patients suffering of gastro-esophageal reflux (GER). However, long term instrumental evaluations of GER after LRYGB are not available.

The aim of this study is to evaluate the long-term effects of laparoscopic Roux-en-Y Gastric Bypass (LRYGB) on gastro-esophageal function.

DETAILED DESCRIPTION:
Consecutive morbidly obese patients selected for LRYGB were included in a prospective study. The investigators performed clinical evaluation with GERD-HRQoL and GIS questionnaire, upper endoscopy, esophageal manometry and 24h-impedance pH monitoring (24h-MII-pH) preoperatively and at 12 and 60 months after surgery. Patients were divided into 2 groups according to the presence of GER at preoperative 24h-MII-pH.

ELIGIBILITY:
Inclusion Criteria:

* history of obesity exceeding 5 years
* documented previous weight loss attempts,
* body mass index (BMI)) of 40-50 kg/m2
* age of 18-60 years.

Exclusion Criteria:

* contraindications to pneumoperitoneum
* large esophageal hiatal hernia
* pregnancy,
* drug or alcohol abuse,
* psychological disorders (e.g., bulimia, depression)
* hormonal or genetic obesity-related disease
* previous gastric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive morbidly obese patients selected for LRYGB
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2006-05; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of weakly acidic reflux | preoperatively, 12 and 60 months after LRYGB
  number of weakly acidic reflux at 24 hour pH impedance monitoring

SECONDARY OUTCOMES:
GERD-HRQoL clinical score | preoperatively, 12 and 60 months after LRYGB
  Standard and previous validated questionnaire was employed in the study to assess gastroesophageal function and quality of life
Lower esophageal sphincter pressure | preoperatively, 12 and 60 months after LRYGB
  Esophageal manometry measures lower esophageal sphincter pressure
Amplitude of esophageal peristaltic waves | preoperatively, 12 and 60 months after LRYGB
  Esophageal manometry evaluates amplitude of esophageal peristalsis
Grade of esophagitis | preoperatively, 12 and 60 months after LRYGB
  Upper endoscopy is performed to assess the presence of esophagitis
Number of acidic reflux | preoperatively, 12 and 60 months after LRYGB
  number of acidic reflux at 24 hour pH impedance monitoring

REFERENCES:
- [Result] Vela MF. Non-acid reflux: detection by multichannel intraluminal impedance and pH, clinical significance and management. Am J Gastroenterol. 2009 Feb;104(2):277-80. doi: 10.1038/ajg.2008.23. No abstract available. PMID 19190606
- [Result] Sundbom M, Hedenstrom H, Gustavsson S. Duodenogastric bile reflux after gastric bypass: a cholescintigraphic study. Dig Dis Sci. 2002 Aug;47(8):1891-6. doi: 10.1023/a:1016429603337. PMID 12184547
- [Result] Collard JM, Romagnoli R. Roux-en-Y jejunal loop and bile reflux. Am J Surg. 2000 Apr;179(4):298-303. doi: 10.1016/s0002-9610(00)00326-3. PMID 10875990
- [Result] Mabrut JY, Collard JM, Romagnoli R, Gutschow C, Salizzoni M. Oesophageal and gastric bile exposure after gastroduodenal surgery with Henley's interposition or a Roux-en-Y loop. Br J Surg. 2004 May;91(5):580-5. doi: 10.1002/bjs.4569. PMID 15122609
- [Result] Barak N, Ehrenpreis ED, Harrison JR, Sitrin MD. Gastro-oesophageal reflux disease in obesity: pathophysiological and therapeutic considerations. Obes Rev. 2002 Feb;3(1):9-15. doi: 10.1046/j.1467-789x.2002.00049.x. PMID 12119661
- [Derived] Rebecchi F, Allaix ME, Ugliono E, Giaccone C, Toppino M, Morino M. Increased Esophageal Exposure to Weakly Acidic Reflux 5 Years After Laparoscopic Roux-en-Y Gastric Bypass. Ann Surg. 2016 Nov;264(5):871-877. doi: 10.1097/SLA.0000000000001775. PMID 27429035